CLINICAL TRIAL: NCT04073459
Title: A Multi-center, Randomized, Active-controlled, Parallel-group, Open-label and Phase II Study to Evaluate Immunogenicity and Safety of LBVD (Fully Liquid Hexavalent Vaccine; Adsorbed Diphtheria-Tetanus-Pertussis-Hepatitis B- Inactivated Poliomyelitis (Sabin) and Haemophilus Influenzae Type b Conjugate Vaccine) Compared to Co-administration of EupentaTM Inj. and Imovax® Polio (Poliomyelitis Vaccine (Inactivated)) in Separate Injections in Healthy Infants at 6-10-14 Weeks of Age as Primary Series
Brief Title: Safety and Immunogenicity of Hexavalent Vaccine(DTwP-HepB-IPV-Hib) in Healthy Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VDCL002
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type b Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- L dose of Hexavalent (Experimental): Low dose of candidate hexavalent vaccine (DTwP-HepB-Sabin IPV-Hib)
  Interventions: Biological: DTwP-HepB-Sabin IPV-Hib
- M dose of Hexavalent (Experimental): Middle dose of candidate hexavalent vaccine (DTwP-HepB-Sabin IPV-Hib)
  Interventions: Biological: DTwP-HepB-Sabin IPV-Hib
- H dose of Hexavalent (Experimental): High dose of candidate hexavalent vaccine (DTwP-HepB-Sabin IPV-Hib).
  Interventions: Biological: DTwP-HepB-Sabin IPV-Hib
- Pentavalent+IPV (Active Comparator): Co-administration of EupentaTM Inj and Imovax Polio
  Interventions: Biological: Pentavalent vaccine and Salk IPV

INTERVENTIONS:
Biological: DTwP-HepB-Sabin IPV-Hib — Intramuscular injection into the anterolateral area of the thigh
  Arms: H dose of Hexavalent; L dose of Hexavalent; M dose of Hexavalent
Biological: Pentavalent vaccine and Salk IPV — Intramuscular injection into anterolateral area of the thigh
  Arms: Pentavalent+IPV

SUMMARY:
The purpose of the study is to evaluate immunogenicity and safety of three different doses of candidate hexvalent vaccine in comparison to co-administration of EupentaTM Inj. and Imovax® Polio in separate injections at four weeks after completion of three-dose primary series at 6-10-14 weeks of age when administered to healthy infants and thereby to select the optimal dose of candidate vaccine

ELIGIBILITY:
Inclusion Criteria:

1. A male or female healthy (i.e. free of obvious health problems) infant who have reached at least 42 days (6 weeks) of age and not more than 56 days (8 weeks) of age at the time of first vaccination
2. Born at full term pregnancy (Gestational age ≥ 37 weeks)
3. Body weight ≥ 3.2 kg at the time of screening
4. Received one dose of hepatitis B mono-vaccine within seven days of birth
5. Born to both hepatitis B virus surface antigen (HBsAg) and human immunodeficiency virus (HIV) negative mother
6. Subject's parent(s) or Legally Acceptable Representative (LAR) able to understand and comply with planned study procedures
7. Written informed consent by subject's parent(s) or LAR

Exclusion Criteria:

1. Previously received any dose of diphtheria, tetanus, pertussis, polio and/or Hib containing vaccines
2. History of previous or concurrent vaccinations other than hepatitis B, Bacillus Calmette-Guerin (BCG), rotavirus and pneumococcal vaccine
3. Known or suspected history of diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, or Hib diseases
4. Household contact and/or intimate exposure in the previous 30 days to an individual with ascertained diphtheria, pertussis, hepatitis B, polio or Hib diseases
5. Experienced fever ≥ 38°C (100.4°F) within the past three days prior to screening
6. Experienced significant acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the past seven days prior to screening
7. Known or suspected immune disorder or immunodeficient condition
8. Receipt of immunoglobulin or blood-derived product since birth
9. Chronic administration (defined as more than 14 days) of immunosuppressant or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone, or equivalent, ≥0.5mg/kg/day. Inhaled and topical steroids are allowed.
10. History of bleeding disorder contraindicating intramuscular injection
11. Major congenital defects or serious chronic illness
12. History of any neurological disorders or seizures
13. History of allergic reactions to any vaccine components including excipients and preservatives (neomycin, streptomycin, polymyxin B, yeast or etc.)
14. History of allergic reactions to latex
15. Participation in another interventional trial or received any investigational product within 30 days before to the enrollment
16. Plan to leave the area of the study site before the end of the study period
17. Infants who are considered unsuitable for the clinical study by the investigator

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
seroprotection/seroconversion/vaccine-response rate | 4 weeks after three-dose primary series
  Proportion of subjects achieving seroprotection/seroconversion/vaccine-response to each antigenic components

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) or Geometric mean titer (GMT) | 4 weeks after three-dose primary series
  GMC or GMT and their ratio of all types of antibodies
Seroprotection rate against diphtheria with cut-off ≥ 1.0 IU/mL | 4 weeks after three-dose primary series
  Proportion of subjects achieving anti-diphtheria toxoid antibody level with cut-off ≥ 1.0 IU/mL
Seroprotection rate against tetanus with cut-off ≥ 1.0 IU/mL | 4 weeks after three-dose primary series
  Proportion of subjects achieving anti-tetanus toxoid antibody level with cut-off ≥ 1.0 IU/mL
Seroprotetion rate against PRP with cut-off ≥ 1 µg/mL | 4 weeks after three-dose primary series
  Proportion of subjects achieving anti-PRP antibody level with cut-off ≥ 1 µg/mL
Seroconversion rate against Salk serotypes | 4 weeks after three-dose primary series
  Proportion of subjects achieving seroconversion of each Salk wild poliovirus serotype
Seroprotection rate against Sabin and Salk serotypes | 4 weeks after three-dose primary series
  Proportion of subjects achieving seroprotection of each Sabin and Salk poliovirus serotype